CLINICAL TRIAL: NCT01513993
Title: RENEWING HEALTH - Large Scale Pilot in Veneto Region: Remote Monitoring of Chronic Heart Failure
Brief Title: Remote Monitoring of Chronic Heart Failure in Veneto Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regione Veneto (Other)
Collaborators: European Commission (Other); Azienda Unità Locale Socio Sanitaria n.9 Treviso (Other); Azienda ULSS 7 Conegliano (Other); Azienda ULSS 16 Padova (Other); Azienda ULSS di Verona e Provincia (Other); Azienda ULSS 12 Veneziana (Other); Azienda Unità Socio Sanitaria di Dolo Mirano (Other); Azienda Ospedaliera di Padova (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: G. A. 250487-Veneto WP8Cl7
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2012-01

CONDITIONS: Congestive Heart Failure
Keywords: CHF; Telemonitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Treatment as usual
- Telemonitoring for patients with Congestive Heart Failure (Experimental)
  Interventions: Procedure: Telemonitoring for patients with Congestive Heart Failure

INTERVENTIONS:
Procedure: Telemonitoring for patients with Congestive Heart Failure — Patients are equipped with a telemonitoring kit composed by a portable wrist-clinic device and digital weight scale for clinical parameters measuring and a gateway device for data transmission.
  The patient can monitor a complete set of clinical parameters, such as pulse-oxymetry, heart rate, blood pressure, ECG and body weight, with a frequency set by the clinician in the personalised treatment plan. Data are transmitted to a regional eHealth centre where a group of operators keeps these information under control and alerts the reference clinician in case of worsening of symptoms.
  Arms: Telemonitoring for patients with Congestive Heart Failure

SUMMARY:
The purpose of this study is to evaluate whether telemonitoring of patients with chronic heart failure produces a reduction in the combined end point of all cause mortality and number of hospitalisations, and whether it improves health related quality of life. In addition, the trials evaluate the economic and organisational impact of the telemonitoring service and examine its acceptability by patients and health professionals.

DETAILED DESCRIPTION:
The study is designed to evaluate the impact of telemonitoring on the management of CHF compared with outpatient usual care. From a clinical point of view, the trial will allow to investigate how telemonitoring contributes to reduct the combined end point of all cause mortality and re-hospitalizations, as well as the other kinds of access to hospital facilities (bed-days, specialistic and ER visits). The trial will examine whether the CHF patients improve their health-related quality of life and reduct the anxiety about health conditions, thanks to the telemonitoring. A cost-effectiveness and cost-utility analysis will be carried out in order to determine if and how telemonitoring helps to limit the healthcare expenditure. The evaluation will deal also with organizational changes and task shift due to telemonitoring introduction and patients and professional perception towards the service.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Discharge from hospital after acute heart failure in the previous 3 months and EF < 40% or EF > 40% plus BNP > 400 (or plus NT-proBNP>1500) during hospitalization

Exclusion Criteria:

* Comorbidities prevalent on CHF with life expectation < 12 months.
* Impossibility or inability to use the equipment and help at home not available.
* Myocardial infarction or percutaneous coronary intervention in the last 3 months or scheduled.
* Coronary artery bypass, valve substitution or correction in the last 6 months.
* Being on waiting list for heart transplantation.
* Being enrolled in other trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 315 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Combined end point of all cause mortality and number of hospitalisations for heart failure | 12 months

SECONDARY OUTCOMES:
Cardiovascular and all-cause mortality | 12 months
Health-Related Quality of Life | 12 months
  Health-Related Quality of Life is assessed by the SF-36 questionnaire
Number of hospitalisations (including rehospitalisations) for all causes and for heart failure | 12 months
Total number of days in hospital | 12 months
Number of specialist visits | 12 months
Number of visits at emergency department for heart failure | 12 months
Anxiety and depression status | 12 months
  Anxiety and depression status is assessed by Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Zoran Olivari, DM, Principal Investigator — Azienda Unità Locale Socio Sanitaria n.9 Treviso
Locations (8):
- Italy (8):
  - Azienda Ospedaliera di Padova - Cardiology Department, Padua, Padova
  - Ospedale Immacolata Concezione - Cardiology Department, Piove di Sacco, Padova
  - Presidio ospedaliero di Conegliano - Department of Cardiology, Conegliano, Treviso
  - Ospedale Ca'Foncello - Pulmonology Department, Treviso, Treviso
  - Ospedale di Mirano - Cardiology Department, Mirano, Venezia
  - Ospedale SS Giovanni e Paolo - Cardiology Department, Venezia, Venezia
  - Ospedale San Fracastoro - Cardiology Department, San Bonifacio, Verona
  - Azienda Ospedaliera Universitaria Integrata di Verona - Geriatric Medicine Department, Verona, Verona

REFERENCES:
- [Background] Scherr D, Kastner P, Kollmann A, Hallas A, Auer J, Krappinger H, Schuchlenz H, Stark G, Grander W, Jakl G, Schreier G, Fruhwald FM; MOBITEL Investigators. Effect of home-based telemonitoring using mobile phone technology on the outcome of heart failure patients after an episode of acute decompensation: randomized controlled trial. J Med Internet Res. 2009 Aug 17;11(3):e34. doi: 10.2196/jmir.1252. PMID 19687005
- [Background] Clark RA, Inglis SC, McAlister FA, Cleland JG, Stewart S. Telemonitoring or structured telephone support programmes for patients with chronic heart failure: systematic review and meta-analysis. BMJ. 2007 May 5;334(7600):942. doi: 10.1136/bmj.39156.536968.55. Epub 2007 Apr 10. PMID 17426062
- [Background] Inglis SC, Clark RA, McAlister FA, Stewart S, Cleland JG. Which components of heart failure programmes are effective? A systematic review and meta-analysis of the outcomes of structured telephone support or telemonitoring as the primary component of chronic heart failure management in 8323 patients: Abridged Cochrane Review. Eur J Heart Fail. 2011 Sep;13(9):1028-40. doi: 10.1093/eurjhf/hfr039. Epub 2011 Jul 6. PMID 21733889
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835
- [Background] Klersy C, De Silvestri A, Gabutti G, Regoli F, Auricchio A. A meta-analysis of remote monitoring of heart failure patients. J Am Coll Cardiol. 2009 Oct 27;54(18):1683-94. doi: 10.1016/j.jacc.2009.08.017. PMID 19850208
- [Background] Inglis SC, Clark RA, McAlister FA, Ball J, Lewinter C, Cullington D, Stewart S, Cleland JG. Structured telephone support or telemonitoring programmes for patients with chronic heart failure. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007228. doi: 10.1002/14651858.CD007228.pub2. PMID 20687083
- See also: The Renewing Health project is partially funded under the ICT Policy Support Programme (ICT PSP) as part of the Competitiveness and Innovation Framework Programme by the European Community — http://www.renewinghealth.eu